CLINICAL TRIAL: NCT05806931
Title: Sequential Combined TAS-102 and Oxaliplatin Alternating With TAS-102 and Irinotecan (Sequential TASOXIRI) With Bevacizumab for Late-Line Metastatic Colorectal Cancer
Brief Title: Sequential TAS-OX Alternating With TAS-IRI Plus Bevacizumab for Late-Line Metastatic Colorectal Cancer
Acronym: SCOTI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Howard S. Hochster, MD, Distinguished Professor of Medicine, Director Clinical Oncology Research, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 072303; Pro2023000358 (Other: Rutgers, The State University of New Jersey)
Record Dates: First submitted 2023-03-23; First posted 2023-04-10 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Colon Cancer; Rectal Cancer
Keywords: Sequential Combined TAS-102; Oxaliplatin; Irinotecan; Late-Line Metastatic Colorectal Cancer; Bevacizumab
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — trifluridine tipiracil drug combination; Oxaliplatin; Irinotecan; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tolerability of TAS-102, oxaliplatin, irinotecan with bevacizumab (Experimental): Each treatment cycle will be fourteen days long. TAS-102 25 mg/m2 will be taken orally twice daily on days 1-5 of each cycle. Oxaliplatin 85 mg/m2 infusion will be given on day one for one cycle alternating with Irinotecan 150 mg/m2 infusion, which will be given on day one the next cycle.
  Interventions: Drug: TAS-102, oxaliplatin, irinotecan with bevacizumab

INTERVENTIONS:
Drug: TAS-102, oxaliplatin, irinotecan with bevacizumab — Participants will be treated with the study drugs until radiological evidence of disease progression or until treatment discontinuation secondary to adverse events. TAS-OX alternating with TAS-IRI (sequential TASOXIRI) with Bevacizumab, in the treatment of mCRC.

SUMMARY:
This study is to evaluate the disease control rate and time to progression of the sequential combination of oxaliplatin with an alternative anti-metabolite Trifluridine/tipiracil hydrochloride mixture, TAS-102,(TAS-OX) as well as irinotecan in combination with TAS-102 oxaliplatin(TAS-OX) + Bevacizumab in late-line metastatic colorectal cancer (mCRC)

DETAILED DESCRIPTION:
This phase II trial will evaluate efficacy of TAS-OX alternating with TAS-IRI (sequential TASOXIRI) with Bevacizumab, in the treatment of mCRC. Participants will be treated with the study drugs until radiological evidence of disease progression or until treatment discontinuation secondary to adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage IV colon cancer (AJCC 7th edition) that has progressed after standard therapy that included 5-FU, irinotecan, oxaliplatin and appropriate antibody therapy. Antibody therapy with bevacizumab and an anti-EGFR antibody, if RAS wild type, should have been given unless medical reasons have precluded their use. Participants who could not tolerate standard agents because of unacceptable, but reversible toxicity necessitating their discontinuation will be allowed to participate.
* Participants who had received adjuvant chemotherapy and had recurrence during or within six months of completion of the adjuvant chemotherapy will be allowed to count the adjuvant therapy as one chemotherapy regimen for advanced disease.
* Progression of disease must be documented on the most recent scan.
* Presence of measurable disease
* RAS mutation and MMR status must be determined (or tissue availability for testing if not already determined).
* Age 18 years or older.
* ECOG performance status 0-1.
* Life expectancy of at least three months.
* Participants with adequate organ function:

  1. Absolute neutrophil count (ANC) > 1.5 x 109/L
  2. Hemoglobin > 9 g/dL
  3. Platelets (PLT) > 70 x 109/L
  4. AST/ALT < 5 x ULN
  5. Albumin within normal limits for institution
* Women who are nursing and discontinue nursing prior to enrollment in the program.
* Ability to take oral medication (i.e., no feeding tube).
* Participant able and willing to comply with study procedures as per protocol.
* Participant able to understand and willing to sign and date the written voluntary informed consent form (ICF) at screening visit prior to any protocol-specific procedures.

Exclusion Criteria:

* Participants who have previously received TAS-102.
* Grade 3 or higher peripheral neuropathy (functional impairment).
* Inability to tolerate irinotecan previously (due to uncontrolled diarrhea)
* There are no specific exclusions for bevacizumab. Bevacizumab should be given unless there are specific contraindications per the treating investigator, which should be stated. If UPC is >1.0 (as above) hold bevacizumab until proteinuria resolves and then start bevacizumab.
* Symptomatic CNS metastases requiring treatment.
* Other active malignancy within the last three years (except for non-melanoma skin cancer or a non-invasive/in situ cancer).
* Pregnancy or breast feeding.
* Current therapy with other investigational agents.
* Active infection with body temperature > 38°C due to infection.
* Major surgery within prior four weeks (the surgical incision should be fully healed prior to drug administration).
* Any anticancer therapy within prior two weeks of first dose of study drug.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to TAS-102.
* Current therapy with other investigational agents or participation in another clinical study or any investigational agent received within prior four weeks.
* Grade 3 or higher hypersensitivity reaction to oxaliplatin or irinotecan, or grade 1-2 hypersensitivity reaction to oxaliplatin not controlled with pre-medication.
* Has unresolved toxicity of greater than or equal to Common Terminology Criteria for Adverse (CTCAE) Grade 2 attributed to any prior therapies (excluding anemia, alopecia, skin pigmentation, and platinum-induced neurotoxicity).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Disease control rate (DCR): | From baseline until the date of first documented progression of disease, as assessed up to 100 months
  Defined as the percentage of patients who have achieved complete response (CR), partial response (PR) and stable disease (SD). The disease control rate will be calculated along with 95% confidence interval. As Simon's two stage design is used in the study, 95% CI will be calculated for the two-stage nature of the study design. Response will be determined by independent radiologists using the RECIST criteria.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, on average up to 100 months
  Progression Free Survival (PFS) Progression will be assessed by a CT scan according to RECIST criteria version 1.1. This criterion will be estimated by the median time based on a Kaplan-Meier method. Patients who have not progressed or died at the time of analysis will be censored at the time of their latest follow-up with clinically stable disease. This includes participants who withdraw consent.
Overall Survival (OS) | From date of randomization until the date of death up to 100 months
  This will be analyzed and plotted using the Kaplan-Meier method.
Overall Response Rate (ORR) | From the date of randomization and measured through the course of study treatment, assessed up to 100 months
  This will be calculated along with 95% confidence interval.
  Response rate is defined as the percentage of subjects with a confirmed complete response (CR) or partial response (PR) by investigator assessment as per RECIST criteria, version 1.1. A maximum of five measurable lesions in total (and up to 2 per organ) representative of all involved organs should be identified as target lesions at baseline and measured through the course of study treatment. At baseline, the sum of the diameters (longest diameters (LD) for extra nodal target lesions and short axis diameters (SAD) for nodal lesions) will be calculated and reported as the baseline sum LD. This baseline sum LD will be used as the reference by which to characterize the objective tumor response. All other lesions should be identified as non-target lesions and should also be recorded at baseline. Measurements of these lesions are not required, but the presence or absence of each should be noted throughout the study
Duration of Response | From the date of response until the date of first documented disease progression or death, assessed up to 100 months
  Response will be determined by independent radiologist using RECIST 1.1. Time to progression for responders will be analyzed by Kaplan-Meier methods.

CONTACTS AND LOCATIONS:
Overall Officials: Howard S. Hochster, MD, Principal Investigator — Cancer Institute of New Jersey Rutgers
Locations (9):
- United States (9):
  - Trinitas Hospital and Comprehensive Cancer Center, Elizabeth, New Jersey
  - RWJBarnabas Health Jersey City Medical Center, Jersey City, New Jersey
  - RWJBarnabas Health - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - Cooperman Barnabas Medical Center (Saint Barnabas Medical Center), Livingston, New Jersey
  - RWJBarnabas Health - Monmouth Medical Center, Long Branch, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - RWJBarnabas Health - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - RWJBarnabas Health - Robert Wood Johnson University Hospital, Somerset, New Jersey
  - RWJBarnabas Health - Community Medical Center, Toms River, New Jersey

IPD SHARING:
Plan to Share IPD: No